CLINICAL TRIAL: NCT06784609
Title: Correlation of Euroscore-II, STS Risk Scoring Systems and Frailty Tests with Cardiac Histopathological Findings in Coronary Bypass Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Zülfiye Yıldız, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: KAEK-11/28.08.2024.133
Record Dates: First submitted 2024-09-06; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Coronary Arterial Disease (CAD); Fraility; Histopathology; Cardiac Risk Factors; Mortality; Morbidities; Coronary Artery Bypass; Anesthesia; Preoperative Cardiac Surgery Patients
Keywords: coronary arterial disease; cad; coronary artery bypass; coronary; fraility; histopathology; cardiac risk factors; mortality; morbidities; bypass; preoperative cardiac surgery patients
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Coronary Artery Bypass Surgery — Coronary Artery Bypass Surgery

SUMMARY:
Various risk classification systems are used to predict postoperative mortality and morbidity development in cardiac surgery. Risk calculation with these systems is a guide in determining preoperative strategies, performing cost analyses, creating different treatment options and classifying diseases according to their severity. In recent years, tests defined as Frailty, which show how independently a person can perform daily living activities and are also associated with postoperative complications, have also been used. These tests allow for a personalized approach such as determining the most appropriate treatment options and pre- and postoperative rehabilitation.

This study aims to evaluate the risk scores used to predict mortality during the preoperative preparation process in cases planned for elective Coronary Artery Bypass Graft (CABG) using the European System for Cardiac Operative Risk Evaluation (Euroscore)-II and Society of Thoracic Surgeons (STS) as well as Frailty with the Katz Index and modified Rockwood Clinical Frailty Scale, and to correlate the findings obtained from the histopathological study of the tissue sample taken from the right atrium during the operation with the test results.

Secondary objectives are to investigate the compatibility of the age-related changes detected histopathologically with chronological age, to reveal which of the Frailty tests used gives better results in predicting mortality, and on the other hand, to reveal the relationship between Frailty tests and STS and Euroscore-II.

DETAILED DESCRIPTION:
Various risk classification systems are used to predict postoperative mortality and morbidity development in cardiac surgery. Risk calculation with these systems is a guide in determining preoperative strategies, performing cost analyses, creating different treatment options and classifying diseases according to their severity. In recent years, tests defined as Frailty, which show how independently a person can perform daily living activities and are also associated with postoperative complications, have also been used. These tests allow for a personalized approach such as determining the most appropriate treatment options and pre- and postoperative rehabilitation.

This study aims to evaluate the risk scores used to predict mortality during the preoperative preparation process in cases planned for elective Coronary Artery Bypass Graft (CABG) using the European System for Cardiac Operative Risk Evaluation (Euroscore)-II and Society of Thoracic Surgeons (STS) as well as Frailty with the Katz Index and modified Rockwood Clinical Frailty Scale, and to correlate the findings obtained from the histopathological study of the tissue sample taken from the right atrium during the operation with the test results.

Secondary objectives are to investigate the compatibility of the age-related changes detected histopathologically with chronological age, to reveal which of the Frailty tests used gives better results in predicting mortality, and on the other hand, to reveal the relationship between Frailty tests and STS and Euroscore-II.

The STS scoring system was developed in 1994 and is a widely used system in the world that allows for the evaluation of morbidity as well as expected mortality for open heart surgery. The Euroscore -II system is also one of the most widely used systems in this field. Both methods are simple, accurate, provable and inexpensive.

In the assessment of frailty, the Clinical Frailty Scale (CFS) was first introduced by Rockwood and colleagues in 2005. This scale was modified by Pulok and colleagues in 2020. CFS is shown to be the most practical method (can be completed in less than a minute) that can also be applied in the field of Emergency Medicine. In 1963, Katz developed the Katz Activities of Daily Living (ADL) Scale, which shows how independently older individuals can perform daily activities. Although frailty is defined as related to aging, it has been accepted as a concept independent of age in recent years.

When evaluated histopathologically, changes such as hypertrophy, fibrosis, protein misfolding, and accumulation of dysfunctional mitochondria have been shown in the aging heart. Age-related changes in the heart are thought to be due to oxidative stress, non-enzymatic glycation, inflammation, and changes in cardiovascular gene expression. Age is a risk factor for the development of many diseases, and it has been shown that frail individuals have a higher susceptibility to disease than healthy individuals of the same age.

The investigators aimed to demonstrate the histopathological prediction degree and corresponding value of risk scores and fragility index values on cardiac tissue and to demonstrate the reality and importance of these scoring systems at the tissue level and to evaluate their reliability in predicting postoperative mortality and morbidity development. In addition, the investigators aimed to reveal the relationship of fragility tests with both age and STS and Euroscore-II by examining the compatibility of age-related changes detected histopathologically with chronological age.

The tests to be used for this study are routine tests and there is no risk. The cardiac tissue to be used for histopathological examination is tissue pieces that are dissected from the right atrial appendage while removing the venous cannula and routinely removed from the body and sent for histopathological examination. Since no non-routine tissue or blood sample will be taken from the patient, there is no risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 40 and 80,
* Under general anesthesia, planned for elective isolated CABG.

Exclusion Criteria:

* Under the age of 40, over the age of 80,
* Emergency cases,
* Reoperations,
* Patients with EF ≤ 25%,
* Patients with vasculitis, rheumatological diseases and connective tissue diseases.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients between the ages of 40 and 80,
  * Under general anesthesia, planned for elective isolated CABG.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Histopathological Examination | Within the following month after the procedure
  Within the scope of histopathological examination; inflammation and fibrosis criteria in cardiac tissue will be evaluated by the Pathologist and will be interpreted by grading as 0, 1, 2, 3.

OTHER OUTCOMES:
Cardiac Risks Scoring Systems | At the first day of enrollment
  Within the scope of STS; laboratory values, preoperative medications, diabetes, endocarditis, illicit drug use, alcohol use, tobacco use, chronic lung disease, vascular diseases and cardiac status will be assessed through the operational risk calculator on the STS website.
  Within the scope of Euroscore -II; chronic lung disease, extracardiac arteriopathy, poor mobility, previous cardiac surgery, active endocarditis, critical preoperative status, renal failure, insulin-using diabetes, cardiac factors and operative factors will be assessed through the calculator on the Euroscore website.
  STS score: Will be presented as percentage (numerical data)
  EUROSCORE 2: Will be presented as percentage (numerical data)
Fraility Tests | At the first day of enrollment
  Within the scope of the Rockwood modified clinical frailty scale (CFR); the patients' vitality and frailty in daily living activities will be evaluated out of 9 points. CFS level 2 "Fit", level 4 "Living with Very Mild Frailty", levels 5-8 are "Living with..." mild, moderate, severe, and very severe frailty, respectively
  Within the scope of the Katz Daily Living Activities Scale (ADL); the extent to which daily activities can be performed independently in elderly individuals will be evaluated out of 6 points.
  Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
  Rockwood scale: Will be presented as level (ordinal data)
  Katz scale: Will be presented as the score they will receive and the group they are included in will be interpreted according to this score (numerical data)

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiye Yildiz M.D., Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No